CLINICAL TRIAL: NCT01889342
Title: Metacognitive Therapy Versus Cognitive Behavioral Therapy for Mixed Anxiety Disorders: A Randomized Controlled Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Modum Bad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SveJoh 1
Record Dates: First submitted 2013-06-26; First posted 2013-06-28 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Mixed Anxiety Disorders
Keywords: MCT; Metacognitive therapy; Anxiety disorders; Transdiagnostic
MeSH Terms: conditions — Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metacognitive therapy (Experimental): The treatment is based on the generic manual by Wells (2009).
  Interventions: Behavioral: Metacognitive therapy
- Cognitive behavorial therapy (Active Comparator): CBT includes the diagnose specific manuals for panic disorder (Clark, 1986), Social Phobia (Clark & Wells, 1995) and PTSD (Foa, 2007).
  Interventions: Behavioral: Cognitive behavioral therapy

INTERVENTIONS:
Behavioral: Metacognitive therapy
  Arms: Metacognitive therapy
Behavioral: Cognitive behavioral therapy
  Arms: Cognitive behavorial therapy

SUMMARY:
Comorbidity is normal in clinical practice. Metacognitive Therapy (MCT) is a transdiagnostic model and could therefore be well suited when it comes to treating patients with high rates of comorbidity. So far, no studies have examined MCT in comparison with the best documented and evidence based treatment, cognitive behavioral treatment(CBT), in a randomized controlled trial consisting of mixed anxiety disorder sample with high degree of comorbidity.

The main aim of this study is to 1) Evaluate the effectiveness of metacognitive therapy in a sample of mixed anxiety disorders as compared to a group receiving existing evidence-based single diagnosis CBT- treatment protocols 2) Investigate patterns and mechanisms of change in the two treatments.

ELIGIBILITY:
Inclusion Criteria:

* DSM IV diagnoses of SAD, PD/A or PTSD (CSR>4)
* Withdraw of all psychotropic medications before treatment

Exclusion Criteria:

* Psychosis
* Not willing to accept randomization
* Comorbid conditions are in immediate need of treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Anxiety Disorders Interview Schedule for DSM-IV-Lifetime Version | PRE/POST/1 year follow up
  The ADIS -IV is a semistructured diagnostic interview designed to establish reliable DSM-IV anxiety, mood, somatoform and substance disorders. Interviewers assign a 0-8 clinical severity rating (CSR), that indicate their judgement of the degree of distress.
Beck Anxiety Inventory (BAI) | PRE/POST/weekly and 1 year follow up

SECONDARY OUTCOMES:
The Symptom Checklist 90(SCL90; Derogatis et al., 1996) | Pre/Post/1 year follow up
The Patient Health Questionnaire depression module (PHQ 9; Spitzer et al., 1999) | Pre/Post and 1 year follow up
Metacognitions Questionnaire- 30 (MCQ-30; Wells & Cartwright-Hatton, 2003) | Pre/Post/weekly and 1 year follow up
Working Alliance Inventory (WAI; Horwath & Greenberg, 1989) | Pre/Post/weekly and 1 year follow up
Cognitive attentional syndrome 1 (CAS1; Wells, 2009) | Pre/Post/weekly and 1 year follow up
The Repetitive Thinking Questionnaire(RTQ; McEvoy et al., 2010) | Pre/Post and 1 year follow up
PTSD Symptom scale Self Report (PSSR; Foa et al., 1993) | Pre/Post and 1 year follow up
Social Phobia Inventory (SPIN; Connor et al., 2000) | Pre/Post and 1 year follow up
Mobility inventory (MI; Chambless, 1985) | Pre/Post and 1 year follow up
SF 36 | Pre/Post and 1 year follow up
The Penn State Worry Questionnaire (PSWQ; Meyer, Miller, Metzger & Borkovec, 1990) | Pre/Post and 1 year follow up
Youngs Schema Questionnaire YSQ -75 (Young, 1998) | Pre/Post and 1 year follow up
The Inventory of Interpersonal Problems (IIP 64 C; Horowitz et al., 1988) | Pre/Post and 1 year follow up
Dysfunctional emotion regulations scale (DERS; Graz & Roemer, 2004) | Pre/Post/ and 1 year follow up

CONTACTS AND LOCATIONS:
Overall Officials: Asle Hoffart, Ph.D, Study Chair — Modum Bad and University of Oslo; Sverre Urnes Johnson, MA, Principal Investigator — Modum Bad and University of Oslo
Locations (1):
- Modum Bad, Vikersund, Buskerud, Norway

REFERENCES:
- [Derived] Johnson SU, Hoffart A, Nordahl HM, Ulvenes PG, Vrabel K, Wampold BE. Metacognition and cognition in inpatient MCT and CBT for comorbid anxiety disorders: A study of within-person effects. J Couns Psychol. 2018 Jan;65(1):86-97. doi: 10.1037/cou0000226. Epub 2017 May 25. PMID 28541060